CLINICAL TRIAL: NCT06619236
Title: A Phase 3 Randomized, Open-label Study of Rinatabart Sesutecan (Rina-S) Versus Treatment of Investigator's Choice (IC) in Patients With Platinum Resistant Ovarian Cancer
Brief Title: Study to Assess the Efficacy of Rina-S Compared to Treatment of Investigator's Choice in Participants With Platinum Resistant Ovarian Cancer
Acronym: RAINFOL-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCT1184-02; jRCT2031250064 (Registry Identifier: jRCT); CTR20253987 (Registry Identifier: ChinaDrugTrials.org.cn); PRO1184-002 (Other: Other Sponsor Identifier); GOG-3107 (Other: Other Sponsor Identifier); ENGOT-OV86 (Other: Other Sponsor Identifier); 2024-514822-21 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2024-09-20; First posted 2024-10-01 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Platinum-resistant Ovarian Cancer
Keywords: antibody-drug conjugate; folate receptor alpha (FRα); ovarian cancer; fallopian tube cancer; primary peritoneal cancer; folate receptor; platinum-resistant ovarian cancer (PROC); rinatabart sesutecan; Topoisomerase 1 inhibitor; PRO1184; GEN1184
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; Topotecan; liposomal doxorubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rina-S (Experimental)
  Interventions: Drug: Rina-S
- Investigator's Choice (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Topotecan; Drug: Pegylated liposomal doxorubicin (PLD); Drug: Gemcitabine

INTERVENTIONS:
Drug: Rina-S — Intravenous (IV) infusion
  Other Names: PRO1184; Rinatabart Sesutecan; GEN1184
  Arms: Rina-S
Drug: Paclitaxel — IV infusion
  Arms: Investigator's Choice
Drug: Topotecan — IV infusion
  Arms: Investigator's Choice
Drug: Pegylated liposomal doxorubicin (PLD) — IV infusion
  Arms: Investigator's Choice
Drug: Gemcitabine — IV infusion
  Arms: Investigator's Choice

SUMMARY:
This phase 3 study will be conducted in different countries all over the world.

The purpose of this study is to compare how well Rina-S works against platinum-resistant ovarian cancer compared to chemotherapy drugs that are already approved and used for platinum-resistant ovarian cancer.

Treatment in this study could be Rina-S or it could be 1 of 4 indicated chemotherapy agents that are considered standard medical care. There is an equal (50:50) chance of getting Rina-S or an approved chemotherapy agent as treatment in this study. No one will know what treatment they are assigned to until the first dose.

All participants will receive active drug; no one will be given placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have histologically or cytologically confirmed high grade serous or endometrioid epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer.
* Participants may be enrolled regardless of FRα expression level.
* Participants must have received 1 to 4 prior lines of therapy. Participants must have progressed radiographically on or after their most recent line of therapy.
* Participants must have received prior treatment with the following therapies:

  * Platinum chemotherapy
  * Prior bevacizumab (or biosimilar) treatment is required, if labeled and available as standard of care per institutional guidelines, unless the participant has a documented contraindication or unless the participant is not eligible for treatment with bevacizumab (or biosimilar) due to precautions/intolerance
  * Participants with known or suspected deleterious germline or somatic breast cancer gene (BRCA) mutations and who achieved a complete or partial response to platinum-based chemotherapy must have been treated with a poly ADP-ribose polymerase (PARP) inhibitor as maintenance treatment unless the participant is not eligible for treatment with PARP inhibitor
  * Mirvetuximab soravtansine, if:

    * Mirvetuximab soravtansine is available in the enrollment region, and
    * The participant is eligible based on positive FRα expression per Food and Drug Administration (FDA)-approved (or local equivalent) test, and
    * The participant does not have a documented medical exception, including chronic corneal disorders, history of corneal transplantation, or active ocular conditions requiring ongoing treatment/monitoring, such as uncontrolled glaucoma, wet age-related macular degeneration requiring intravitreal injections, active diabetic retinopathy with macular edema, macular degeneration, presence of papilledema, and /or monocular vision.
* Participants must have platinum-resistant disease:

  * Participants who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum therapy, and must have either had a response (CR or PR) or had non-measurable disease at the start of adjuvant platinum-based therapy, and then progressed between > 91 days and ≤ 183 days after the date of the last dose of platinum.
  * Participants who have received 2 to 4 lines of platinum-based therapy must have progressed on or within 183 days after the date of the last dose of platinum.

Key Exclusion Criteria:

* Prior therapy with an antibody-drug conjugate containing a topoisomerase 1 inhibitor.
* Have primary platinum-refractory disease, defined as ovarian cancer that did not respond (CR or PR) to or progressed ≤ 91 days after the last dose of a first-line platinum-containing regimen.
* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death (e.g., 5-year OS ≥90%), including, but not limited to, adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, ductal carcinoma in situ, or Stage I uterine cancer.
* Known active central nervous system metastases or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry after brain metastasis treatment, they have no new or enlarging brain metastases, and are off corticosteroids and anticonvulsants prescribed for symptoms associated with brain metastases for at least 7 days prior to the first dose of study drug. Participants with suspected brain metastases at screening should undergo a computed tomography (CT)/magnetic resonance imaging (MRI) of the brain prior to study entry.
* Hospitalization or clinical symptoms due to gastrointestinal obstruction within the past 91 days or radiographic evidence of gastrointestinal obstruction at the time of screening. Enrollment of participants who currently require parenteral nutrition must be discussed with the study medical monitor to determine eligibility.
* Ascites requiring frequent paracentesis (more often than approximately every 4 weeks) for symptomatic management. Enrollment of participants with an indwelling peritoneal catheter must be discussed with the medical monitor to determine eligibility.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death (PD) due to any cause, whichever occurs first based on response evaluation criteria in solid tumors (RECIST) version 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 3 years
  OS is defined as the time from date of randomization to date of death due to any cause.
Objective Response Rate (ORR) | Up to approximately 3 years
  ORR is defined as the percentage of participants with best overall response (BOR) of complete response (CR) or partial response (PR) based on RECIST v1.1 as assessed by the investigator.
PFS as Determined by BICR | Up to approximately 3 years
  PFS is defined as the time from the date of randomization to the date of the first documented progression or death (PD) due to any cause, whichever occurs first based on RECIST version 1.1 as determined by BICR.
ORR as Determined by BICR | Up to approximately 3 years
  ORR is defined as the percentage of participants with BOR of CR or PR based on RECIST v1.1 as determined by BICR.
Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from the onset date of response to the date of the first documented progression or death due to any cause based on RECIST v1.1 as assessed by the investigator and by blinded independent central review (BICR).
Percentage of Participants Who Achieved Cancer Antigen-125 (CA-125) Response per Gynecologic Cancer Intergroup (GCIG) Criteria | Up to approximately 3 years
  A CA-125 response per the GCIG criteria is defined as a ≥ 50% reduction in CA-125 levels from baseline.
Time to Second Disease Progression or Death From any Cause (PFS2) | Up to approximately 3 years
  PFS2 is defined as the time from randomization to the date of the second PD (i.e., the first PD reported in subsequent anti-cancer therapies, or long-term follow up) or death.
Overall Change From Baseline in Global Health Status/Quality of Life (GHS/Qol) | Baseline, up to approximately 3 years
  Overall change from baseline in GHS/Qol score (items 29 and 30) will be calculated using the European Organization for Research and Treatment of Cancer Quality of Life Core 30 (EORTC-QLQ-C30) questionnaire. The score ranges from 0 to 100. A high scale score represents a higher response level.
Time to Deterioration (TTD) in the GHS/Qol Score | Up to approximately 3 years
  TTD in the GHS/Qol score is defined as the time from baseline to the first onset of a ≥10-point negative change (decrease) in GHS/QoL score. A longer TTD indicates a better outcome.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to approximately 3 years
Change from Baseline in Electrocardiogram (ECG) Findings to Assess Changes in QTc Associated with Rina-S by Holter Monitor | Baseline through Cycle 3 (Cycle length=21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (175):
- United States (72):
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Arizona Center for Cancer Care (ACCC) - Biltmore, Scottsdale, Arizona
  - University of Arizona Cancer Center - Research and Administration at Main Campus, Tucson, Arizona
  - Providence Saint Joseph Medical Center - Roy and Patricia Disney Family Cancer Center, Burbank, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - USCF Mission Bay, San Francisco, California
  - Kaiser Permanente - Vallejo Medical Center, Vallejo, California
  - UCHealth Cancer Care - Anschutz Medical Campus - University of Colorado Cancer Center, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale School of Medicine, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - SCRI - Florida Cancer Specialists - South Region Research Office, Fort Myers, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Orlando Health Cancer Institute - Downtown Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach, West Palm Beach, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Atlanta, Atlanta, Georgia
  - Augusta University Georgia Cancer Center, Augusta, Georgia
  - Kapi'olani Medical Center for Women and Children, Honolulu, Hawaii
  - Northwest Cancer Center - Dyer, Dyer, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - HCA Midwest Health, Overland Park, Kansas
  - St. Elizabeth Healthcare - Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Louisiana State University Health Sciences Center (LSU Health) - New Orleans, New Orleans, Louisiana
  - Trials365, LLC (Gynecologic Oncology Associates-Shreveport), Shreveport, Louisiana
  - Maine Medical Center Cancer Institute- Scarborough, Scarborough, Maine
  - Holy Cross Health - Holy Cross Hospital, Silver Spring, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health (Spectrum Health), Grand Rapids, Michigan
  - Saint Joseph Mercy Ann Arbor Hospital, Ypsilanti, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Center of Hope, Reno, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Perlmutter Cancer Center - 38th Street, New York, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - New York-Presbyterian - Weill Cornell Medical Center, New York, New York
  - James P. Wilmot Cancer Center, Rochester, New York
  - Duke Cancer Institute, Durham, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - JamesCare Gynecologic Oncology at Mill Run, Hilliard, Ohio
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - USOR - Northwest Cancer Specialists, P.C. dba Compass Oncology - Rose Quarter Cancer Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Health Network - West Penn Hospital, Pittsburgh, Pennsylvania
  - Jefferson Health - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - SCRI Oncology Partners, Nashville, Tennessee
  - USOR - Texas Oncology - Dallas Fort Worth (DFW) - Abilene, Abilene, Texas
  - USOR - Texas Oncology - Dallas Fort Worth (DFW) - Austin Central, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - USOR - Texas Oncology - Dallas Fort Worth (DFW) - Fort Worth, Fort Worth, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - USOR - Virginia Oncology Associates - Norfolk, Norfolk, Virginia
  - Kadlec Clinic - Hematology and Oncology, Kennewick, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University Cancer Institute, Morgantown, West Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- Australia (4):
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Icon Cancer Centre, South Brisbane, Queensland (qld)
  - Mater Misericordiae - Mater Hospital Brisbane, South Brisbane
  - Saint John of God - Subiaco Hospital, Subiaco
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Ordensklinikum Linz GmbH Barmherzige Schwestern, Linz, Upper Austria (Oberösterreich)
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Wien, Vienna
- Belgium (7):
  - Algemeen Ziekenhuis Turnhout - Campus Sint-Elisabeth, Turnhout, Antwerp
  - AZORG - Onze-Lieve-Vrouwziekenhuis - Campus Aalst, Aalst
  - Centre Hospitalier Universitaire Saint-Pierre, Brussels
  - Grand Hôpital de Charleroi - Site Les Viviers, Charleroi
  - Universitair Ziekenhuis (UZ) Leuven - Campus Gasthuisberg, Leuven
  - Centre Hospitalier Chretien - Clinique MontLégia, Liège
  - Algemeen Ziekenhuis Delta - Campus Rumbeke, Roeselare
- Canada (3):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Sunnybrook Health Sciences Centre - Bayview Campus, Toronto
- China (6):
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Hospital of Jilin University, Changchun
  - Zhejiang Cancer Hospital, Hanzhou
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Henan Cancer Hospital - Zhengzhou University, Zhengzhou
- Czechia (7):
  - University Hospital Královské Vinohrady, Prague, Prague
  - Masaryk Memorial Cancer Institute, Brno
  - Fakultní Nemocnice Hradec Králové, Hradec Králové
  - Nemocnice AGEL Nový Jičín a.s., Nový Jičín
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Fakultni nemocnice v Motole, Prague
  - Bulovka University Hospital, Prague
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - The Royal Hospital (Rigshospitalet), Copenhagen
  - Odense Universitets Hospital, Odense
- France (7):
  - Centre Antoine Lacassagne, Nice
  - Hôpital Européen Georges-Pompidou, Paris
  - Hospital Lyon-Sud (HCL), Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Western Cancer Institute - Saint-Herblain - René Gauducheau Site, Saint-Herblain
  - Institut Universitaire du Cancer de Toulouse (IUCT) Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (14):
  - Helios Klinikum Berlin-Buch, Berlin
  - University Hospital Bonn, Bonn
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - University Hospital of Düsseldorf, Düsseldorf
  - Kliniken Essen-Mitte - Evangelische Huyssens-Stiftung, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - Universitätsklinikum Gießen und Marburg - Gießen (UKGM), Giessen
  - Mammazentrum Hamburg am Krankenhaus Jerusalem, Hamburg
  - MVZ Onko Medical GmbH Hanover, Hanover
  - University Hospital Heidelberg /Universitätsklinikum Heidelberg, Heidelberg
  - UniversitY Hospital of Saarland, Homburg
  - Red Cross Hospital Munich, Munich
  - Universitätsklinikum Münster/University Clinic Muenster, Münster
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
- Greece (4):
  - General Hospital of Athens, Athens
  - Attikon University General Hospital/General Hospital of West Attica, Chaïdári
  - Aretaieio Hospital, Léfkos
  - Saint Luke's Hospital, Panórama
- Italy (7):
  - Azienda Sanitaria Locale Brindisi, Brindisi, Apulia
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia/ European Institute of Oncology, Milan
  - Humanitas San Pio X, Milan
  - Local Health Authority of Biella - Nuovo Ospedale degli Infermi, Ponderano
  - Agostino Gemelli University Hospital Foundation IRCCS, Roma
  - Centre Antoine Lacassagne/Azienda Ospedaliera Ordine Mau, Torino
- Japan (14):
  - Aichi Cancer Center, Nagoya, Aichi Pref
  - Kurume University Hospital, Kurume, Fukuoka Pref
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - St. Marianna University Hospital, Kawasaki, Kanagawa Pref
  - Tohoku University Hospital, Sendai, Miyagi Pref
  - Niigata University Medical and Dental Hospital, Niigata, Niigata Pref
  - Okayama University Hospital, Okayama, Okayama Pref.
  - Saitama Medical University - International Medical Center, Hidaka, Saitama Pref.
  - Shizuoka Cancer Center, Nagaizumi-chō, Shizuoka Pref.
  - Jichi Medical University Hospital, Saitama, Tochigi Pref.
  - The Jikei University Hospital, Minato, Tokyo
  - Ehime University Hospital, Shibukawa, Toon City, Ehime Pref
  - National Cancer Center Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
- Netherlands (5):
  - Amsterdam UMC, location VUmc, Amsterdam
  - Medisch Spectrum Twente - Enschede Koningsplein, Enschede
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Maastricht (UMC) Universitair Medisch Centrum, Maastricht
  - Erasmus MC/ Erasmus Medisch Centrum, Rotterdam
- Norway (2):
  - Oslo Universitetssykehus - Radiumhospitalet, Oslo
  - University Hospital of North Norway/Universitetssykehuset Nord-Norge - Tromsø, Tromsø
- Poland (7):
  - Jagiellońskie Centrum Innowacj, Krakow, Lesser Poland (Małopolskie)
  - Białostockie Centrum Onkologii im. Marii Skłodowskiej- Curie w Białymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne w Gdańsku, Gdansk
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Wielkopolskie Centrum Onkologii im. Marii Sklodowskiej-Curie, Poznan
  - Mazowiecki Szpital Wojewódzki im. św. Jana Pawła II w Siedlcach, Siedlce
  - Uniwersytecki Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
- UPR Comprehensive Cancer Center Hospital, Monacillo, San Juan, Puerto Rico
- Spain (8):
  - Hospital Universitario de A Coruña, A Coruña
  - Hospital Universitario DE Donostia, Donostia / San Sebastian
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario La Paz, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Virgen del Rocío University Hospital, Seville
  - IVO - Valencian Institute of Oncology Foundation, Valencia
  - Miguel Servet Hospital, Zaragoza

IPD SHARING:
Plan to Share IPD: No